CLINICAL TRIAL: NCT02406404
Title: Change of Pulmonary Function After Incentive Spirometer Training in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1-2013-0031
Record Dates: First submitted 2015-03-29; First posted 2015-04-02 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2016-03

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- spirometer training group (Experimental): incentive spirometer training group
  Interventions: Behavioral: Incentive spirometer training
- No intervention group (No Intervention): no intervention group

INTERVENTIONS:
Behavioral: Incentive spirometer training — The incentive spirometer, a device that can help improve breathing and strengthen inspiratory muscles. First, the subjects exhaled normally, then placed the mouthpiece in their mouth and sealed their lips around the mouthpiece. Then they inhaled slowly and deeply with their lips sealed tightly on the mouthpiece. After they inhaled as deeply as possible, held their breath for at least 3 seconds, and then removed the mouthpiece from their mouth and breathed out normally. Subjects repeated this technique 10-15 times. When they finished 10-15 exercises, they took a deep breath and coughed. The training was performed ten sessions daily, for 4 weeks.
  Other Names: exercise
  Arms: spirometer training group

SUMMARY:
This study was designed to examine the effect of incentive spirometry in pulmonary rehabilitation of children with cerebral palsy. The incentive spirometer, a device that can help improve breathing and strengthen inspiratory muscles. If the patient assigned to training group, the subjects started to respiratory muscle strengthening exercise using incentive spirometry. The training was performed ten sessions daily, for 4 weeks. Respiratory function tests including forced vital capacity, forced expiratory volume in 1 second, Peak cough flow, maximal phonation time were compared before interventions and at the end of exercise.

ELIGIBILITY:
Inclusion Criteria:

* male or female, 4 to 18 years
* patients who are committed to comply with protocol-required procedures
* GMFCS (Gross motor function classification system) level II, III, IV
* Stable medical condition in the investigator's opinion
* Acceptable chest radiologic result who has no evidence of pulmonary disease

Exclusion Criteria:

* Any uncontrolled clinically significant medical condition other than the one under study
* Patients with cognitive impairment who are unable to comply with protocol-required procedure
* Patients with presence or history of tracheostomy
* Patients who are taking medications that can affect respiratory function

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2013-07; Primary Completion 2015-11-20 (Actual); Study Completion 2015-11-20 (Actual)

PRIMARY OUTCOMES:
Forced vital capacity | within 3 days after respiratory muscle training
  Forced vital capacity means amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Measuring FVC is done through spirometry testing.

SECONDARY OUTCOMES:
forced expiratory volume in 1 second | within 3 days after respiratory muscle training
Peak cough flow | within 3 days after respiratory muscle training
maximal phonation time | within 3 days after respiratory muscle training

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea